CLINICAL TRIAL: NCT06602141
Title: Assessments of Adipogenesis, Lipid Turnover and Cellular Composition in Adipose Tissue in Response to Endurance Exercise
Acronym: ATLAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1805407
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose Clamp Technique; Exercise

STUDY DESIGN:
Masking Description: Participants will be randomized into either the control (CTRL) group or the endurance exercise (EX) group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (CTRL) group (Active Comparator)
  Interventions: Procedure: Muscle Biopsy; Procedure: Adipose Biopsy; Other: Glucose Clamp; Other: Accelerometer; Other: Physical activity/ dietary habits; Other: Heavy Water Labeling Period
- Endurance exercise (EX) group (Active Comparator)
  Interventions: Procedure: Muscle Biopsy; Procedure: Adipose Biopsy; Other: Glucose Clamp; Other: Accelerometer; Other: Endurance Exercise; Other: Heavy Water Labeling Period

INTERVENTIONS:
Procedure: Muscle Biopsy — This procedure is used to sample muscle cells from the leg Vastus Lateralis (thigh) muscle.
Procedure: Adipose Biopsy — This procedure is used to sample fat tissue from the abdomen (belly).
Other: Glucose Clamp — In this test, we will measure the effect of insulin by giving you insulin and glucose (sugar) intravenously through an IV line in your arm.
Other: Accelerometer — The tri-axial accelerometer measure activity and uses those values to estimate the number of calories burned based on your height, weight, age, and gender. The monitor also evaluates physical effort and the body's response to different activities.
Other: Endurance Exercise — Visit the study site 3 times a week to engage in endurance exercise training for approximately 12 weeks. Each session will last approximately 75 minutes, and exercise group can choose to use either a stationary bike or a treadmill to complete the training.
  Arms: Endurance exercise (EX) group
Other: Physical activity/ dietary habits — Visit the study site bi-weekly to get weight measurements and speak to the study team about weight maintenance and participant physical activity/dietary habits.
  Arms: Control (CTRL) group
Other: Heavy Water Labeling Period — Participants in both control groups will be required to drink heavy water, which is ordinary water that is enriched with deuterium (stable, non-radioactive isotope) and called deuterium-labeled water, for 12 weeks.

SUMMARY:
The purpose of this research study is to study the effects of endurance exercise training on adipose (fat) tissue quality and insulin sensitivity in men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Men and pre-menopausal women;
2. 18-45 years of age;
3. BMI 30.0-40.0 kg/m2;
4. For women, if not using pharmaceutical (hormonal) contraception (i.e. birth control pills, vaginal ring, injections, or implant), must agree to use either a double barrier method as a form of birth control to prevent pregnancy (i.e. male condom with spermicide, with or without cervical cap or diaphragm); use implants or intrauterine contraceptive devices; have a tubal ligation (surgically sterile); practice abstinence; or be in an established relationship with a vasectomized or same sex partner during the entire duration of the study;
5. Able to speak and understand written and spoken English;
6. Sedentary defined as self-reporting no more than 1 day per week, lasting no more than 60 minutes, of regular (structured) endurance or resistance exercise in the past year.
7. Must be willing to be randomized to either study group;
8. Must be willing to adhere to all study procedures.
9. Participant has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.

Exclusion Criteria:

1. Self-reported unstable body weight in the last 3 months (> ±5%);
2. Significant changes in the quality of the diet or the level of physical activity within the last 3 months;
3. Weight >396 lb (180 kg);
4. Diagnosis of Type 1 or Type 2 diabetes mellitus;
5. Fasting blood glucose ≥126 mg/dL;
6. HbA1c ≥ 6.5%
7. Blood pressure >140/90 mmHg ;
8. Self-reported history or presence of the following cardiovascular conditions: congestive heart failure, coronary artery disease, significant valvular disease, congenital heart disease, serious arrhythmia, stroke, symptomatic peripheral artery disease, stable angina, myocardial infarction or coronary revascularization within 6 months; clinically significant abnormalities on ECG, presence of cardiac pacemaker, or implanted cardiac defibrillator; inability to complete the VO2max test;
9. Anemia (hemoglobin <12 g/dl in men or 11 g/dl in women; Hct <34%);
10. Kidney disease (creatinine >1.6 mg/dl or estimated glomerular filtration rate <60 mL/min/1.73m2);
11. Abnormal liver enzymes (>2 times the upper limit of normal) that are clinically significant;
12. Serious digestive disorders including severe gastroesophageal reflux disease (GERD), irritable bowel syndrome (IBS), Crohn's disease, chronic constipation and/or diarrhea, etc.;
13. Self-reported chronic, active, or latent infection requiring chronic antibiotic or anti-viral treatment; Human Immunodeficiency Virus (HIV); active hepatitis B or C undergoing antiviral therapy;
14. Current or history of eating disorders;
15. Abnormal bleeding or coagulopathy (self-report) or history of a bleeding disorder or clotting abnormality;
16. Clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD);
17. Dyslipidemia (fasting triglycerides >500 mg/dL; low-density lipoprotein cholesterol (LDL-C) >190 mg/dL);
18. Whole blood donation in the last 3 months or platelet/plasma donation in the last week or plans for donation during entire protocol period;
19. Receiving active treatment (including monoclonal antibodies) for autoimmune disorders within the last 6 months;
20. Alcohol consumption >7 drinks per week for women or 14 drinks per week for men or history of binge drinking (≥5 drinks for males or 4 drinks for females in a 2-hour period more than once per month);
21. Current smokers (smoking or use of any tobacco or e-cigarette/e-nicotine/THC/cannabis products in the last 3 months); stopped smoking <10 years at time of screening for those with a >20 pack-year smoking history or stopped smoking <5 years at time of screening for those with a <20 pack-year smoking history;
22. Night shift work in the last 6 months or planning night shift work during the study period;
23. Known allergy to lidocaine or other local anesthetic;
24. Hyperthyroidism including those with normal TSH (0.35-4.5) on pharmacological treatment; individuals with hypothyroidism may be referred to their primary care provider for evaluation and retested; any medication change for hypothyroidism must be stable for ≥3 months prior to retesting;
25. Previous bariatric or other surgery for obesity;
26. History of cancer (other than non-melanoma skin cancer) within the last 5 years (not in remission); anti-hormonal therapy (e.g., for breast or prostate cancer) within the last 6 months;
27. Diagnosed psychotic or psychiatric conditions prohibiting adherence to study protocol; hospitalization for any psychotic or psychiatric condition within one year;
28. Currently pregnant (pregnancy test performed on day of DEXA scan in women of child-bearing potential); post-partum during the last 12 months; lactating during the last 12 months; planning to become pregnant during the participation period;
29. Polycystic Ovarian Syndrome (PCOS) (self-report);
30. Metabolic bone disease (self-report) including history of non-traumatic fracture from a standing height or less and/or current pharmacologic treatment for low bone mass or osteoporosis, other than calcium, vitamin D, or estrogen;
31. Hospitalization for COVID-19 infection in the past 12 months; individuals who tested positive for COVID-19 but were not hospitalized must be symptom-free at least 14 days;
32. Partial and/or full hysterectomy (self-report);
33. Not willing to archive biospecimens for future use;
34. Not willing to undergo the microdialysis procedure;
35. Participants who fulfill any of the contraindications for MRI including metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos;
36. Unable to participate in MR assessments due to claustrophobia or physical limitations of equipment tolerances (e.g., MRI bore size) based on investigator's judgment at screening;
37. Positive toxicology result from screening;
38. The following medication use is exclusionary:

    * Dose change for any chronic-use drug in the last 3 months;
    * Cardiovascular: beta blockers and centrally acting anti-hypertensive drugs, anticoagulants, antiarrhythmics, and antiplatelet drugs (other than aspirin ≤100 mg/day);
    * Psychiatric: chronic use of medium- or long-acting sedatives and hypnotics, including all benzodiazepines (short-acting non-benzodiazepine sedative-hypnotics are allowed), mood stabilizers, antiepileptic drugs, stimulants, Attention-Deficit/Hyperactivity Disorder (ADHD) drugs, anti-psychotic drugs;
    * Pulmonary/Inflammation: chronic oral steroids (inhaled steroids are allowed), burst/taper oral steroids more than once in the last 12 months, B2-agonists (allowed if on stable dose at least 3 months);
    * Genitourinary: 5-alpha reductase inhibitors, daily phosphodiesterase type 5 inhibitor;
    * Hormonal: androgenic anabolic steroids, anti-estrogens, anti-androgens, estrogens and/or progestins used for reasons other than birth control, growth hormone, insulin like growth factor-I, growth hormone releasing hormone, any drugs used to treat diabetes mellitus or lower blood glucose, metformin for any indication, any drugs used specifically to induce weight loss, any drugs used specifically to induce muscle growth/hypertrophy or augment exercise-induced muscle hypertrophy;
    * Pain/Inflammation: narcotics and narcotic receptor agonists, regular use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen, muscle relaxants ≥2 days per week;
    * Other: chronic systemic antimicrobials (antibiotic, antiviral, antifungal, antiparasite, etc.) for any reason, high-potency topical steroids if ≥10% surface area using rule of 9s, continuous/chronic use of antibiotics or other anti-infectives for treatment or prevention, monoclonal antibodies, anti-rejection medications/immune suppressants;
39. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
In vivo adipogenesis | Before and following 12 weeks of deuterium (2H) labelled water administration and either endurance exercise training or control (no exercise)
  A subcutaneous white adipose tissue biopsy from the abdomen will be collected before and after 12 weeks of deuterium (2H) labelled water administration and either endurance exercise training or control (no exercise). New adipocyte formation will be assessed on frozen isolated 2H2O labelled adipose tissue cells

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Sparks, PhD, Principal Investigator — AdventHealth Translational Research Institute; Ursula White, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - AdventHealth Translational Research Institute, Orlando, Florida
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

REFERENCES:
- See also: AdventHealth Translational Research Institute website — https://www.adventhealthresearchinstitute.com/research/translational-research

DOCUMENTS (1):
  • Study Protocol (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT06602141/Prot_000.pdf